CLINICAL TRIAL: NCT02250950
Title: Decreasing Disparities in Physical Activity: An Intervention Based on Self-Determination Theory and Motivational Interviewing
Brief Title: An Examination of the Efficacy of a Self-Determination Theory and Motivational Interviewing Exercise Intervention
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Syracuse University (Other)
Responsible Party: Principal Investigator, Lauren Miller, Doctoral Candidate, Syracuse University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 4636
Record Dates: First submitted 2014-09-24; First posted 2014-09-26 (Estimated); Last update posted 2015-05-19 (Estimated); Status verified 2015-05

CONDITIONS: Exercise Promotion
Keywords: self-determination theory; motivational interviewing; exercise; physical activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MI and SDT Exercise Group (Experimental): Intervention Condition: Participated in 12 weekly meetings led by MI- and SDT-trained exercise instructor.
  Interventions: Behavioral: MI and SDT Exercise Group
- Non-MI and SDT Exercise Group (Sham Comparator): Control Condition: Participated in 12 weekly meetings led by an exercise instructor who was not trained in MI and SDT.
  Interventions: Behavioral: Non-MI and SDT Exercise Group

INTERVENTIONS:
Behavioral: MI and SDT Exercise Group — The intervention group will participate in a group exercise class that will be held once a week for an hour. This class will be taught by an instructor trained in MI and SDT. This individual will lead group discussions and will have the participants exercise together.
  Arms: MI and SDT Exercise Group
Behavioral: Non-MI and SDT Exercise Group — This group will participate in a group exercise class that will be held once a week for an hour. This class will be taught by an instructor who was not trained in MI and SDT. This individual will lead a regular exercise class.
  Arms: Non-MI and SDT Exercise Group

SUMMARY:
The current study involves conducting an intervention based on self-determination theory (SDT) and motivational interviewing (MI) to promote physical activity in a racially-diverse sample. It is expected that this intervention will successfully increase physical activity in participants.

DETAILED DESCRIPTION:
The mental and physical benefits of physical activity are well-established. However, there is a racial disparity in exercise, such that minorities are much less likely to engage in physical activity than are white individuals. Research suggests that a lack of motivation may be an important barrier to physical activity for racial minorities. Therefore, interventions which increase participants' motivation may be especially useful in promoting physical activity within these groups. A previous meta-analysis has found that physical activity interventions based on self-determination theory (SDT) and motivational interviewing (MI) are especially effective in increasing white individuals' physical activity (Miller & Gramzow, under review). However, it remains unclear the extent to which these results apply to minority populations. The current study involves conducting an intervention based on SDT and MI to promote physical activity in a racially-diverse sample. It is expected that this intervention will successfully increase physical activity in participants. Specifically, it is expected that there will be a greater relative increase in physical activity in minority individuals than white individuals within the intervention group because it is expected that their level of activity will be lower at baseline.

ELIGIBILITY:
Inclusion Criteria:

* participants were were willing to attend an exercise class once a week for 12 weeks, were willing to complete questionnaires at baseline and 12 weeks, allowed the intervention staff to monitor their attendance at the YMCA for 6 months post intervention, and allowed the exercise instructor to create an audio recording of all of the intervention sessions.

Exclusion Criteria:

* not have any illnesses that would prevent them from exercising once a week, not be pregnant or planning to get pregnant within the next 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2014-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
International Physical Activity Questionnaire | 12 weeks

SECONDARY OUTCOMES:
Psychological General Well-Being Index | 12 weeks
Basic Psychological Needs in Exercise Scale | 12 weeks
Behavioural Regulation in Exercise Questionnaire | 12 weeks
Physical Activity Adherence | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lauren S Miller, M.S., Principal Investigator — Syracuse University
Locations (1):
- Lauren S. Miller, Guilderland, New York, United States

REFERENCES:
- [Derived] Miller LS, Gramzow RH. A self-determination theory and motivational interviewing intervention to decrease racial/ethnic disparities in physical activity: rationale and design. BMC Public Health. 2016 Aug 11;16(1):768. doi: 10.1186/s12889-016-3413-2. PMID 27515173